CLINICAL TRIAL: NCT02523287
Title: Clinical Study to Generate a Set of Data Characterising Clinical Events, Physiological Responses, and Innate and Adaptive Immune Responses Following a Single IM Immunisation With Fluad Seasonal Influenza Vaccine or Placebo in Healthy Adults
Brief Title: Placebo Controlled Study to Generate Data Characterising Clinical Events, Physiological Responses and Immune Responses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University of Surrey (Other); Novartis Vaccines (Industry); Max Planck Institute for Infection Biology (Other); deCODE genetics (Industry); VisMederi srl (Industry); GlaxoSmithKline (Industry); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BioVacSafe - Fluad
Record Dates: First submitted 2015-06-24; First posted 2015-08-14 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Safety Markers of Adjuvanted Influenza Vaccine
MeSH Terms: interventions — fluad vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluad - 5 study visits (114 subjects) (Active Comparator): 0,5 ml adjuvanted, subunit seasonal trivalent influenza vaccine (2014-2015). Administration: Intramuscular, deltoid.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 21 (blood sampling).
  Interventions: Biological: Fluad
- Fluad - 3 study visits (114 subjects) (Active Comparator): 0,5 ml adjuvanted, subunit seasonal trivalent influenza vaccine (2014-2015). Administration: Intramuscular, deltoid.
  3 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 7 (blood sampling). On day 21 there's a phone call for safety follow-up.
  Interventions: Biological: Fluad
- Saline - 5 study visits (6 subjects) (Placebo Comparator): 0,5 ml saline. Administration: Intramuscular, deltoid.
  5 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 3 (blood sampling), Day 7 (blood sampling), Day 21 (blood sampling).
  Interventions: Biological: Saline
- Saline - 3 study visits (6 subjects) (Placebo Comparator): 0,5 ml saline. Administration: Intramuscular, deltoid.
  3 out-patient visits: Day 0 (blood sampling, vaccination), Day 1 (blood sampling), Day 7 (blood sampling). On day 21 there's a phone call for safety follow-up.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Fluad — Randomized assignment
  Arms: Fluad - 3 study visits (114 subjects); Fluad - 5 study visits (114 subjects)
Biological: Saline — Randomized assignment
  Arms: Saline - 3 study visits (6 subjects); Saline - 5 study visits (6 subjects)

SUMMARY:
The purpose of this protocol is to generate a set of data that will be analysed by integrated systems biology approach, for validation in subsequent clinical trials or in animal models.

240 healthy participants (18-45y) will be enrolled, 228 will be administered a dose of Fluad on Day 0, 12 will receive a placebo on Day 0.

DETAILED DESCRIPTION:
This study is part of the BIOVACSAFE project, a 5-year project funded by the Innovative Medicine Initiative, which will undertake a series of correlated clinical studies that will apply and develop technologies to generate clinical data on inflammation with licensed vaccines as benchmarks, and identify biomarkers to predict acceptable reactogenicity, for correlation with standardized clinical readouts and inflammatory markers assessed in natural infections.

The purpose of this protocol is to generate a set of data that will be analysed by integrated systems biology approach, for validation in subsequent clinical trials or in animal models. The dataset will broadly characterise:

1. Physiological responses at various time points after immunisation by measuring:

   1. Local and systemic vaccine-related clinical events.
   2. Physiological assessments: heart rate, temperature, blood pressure.
   3. Haematology (blood counts and ESR), biochemistry parameters.
2. Metabolic, innate and adaptive immune responses including:

   1. Innate immune activation detected by global gene expression in whole blood
   2. Metabolic responses detected by metabolic gene expression and pathway activation in whole blood
   3. Adaptive immunity determined by:

   i. Humoral immune response via serum anti-influenza HAI titre

   ii. Cellular immune response via enumeration of HA-specific CD4+ T cells expressing activation markers and/or cytokines following in vitro stimulation and analysis by flow cytometry.

   d. Innate and adaptive immune activation detected by gene pathway activation in whole blood

   e. Immune activation detected by concentration of selected inflammatory soluble mediators in serum including:

   i. chemokines and cytokines

   ii. acute phase proteins
3. Genetic testing of subjects when deemed necessary (genetic testing analysis may be SNIP analysis or full genome analysis).
4. Correlations in changes in innate and adaptive immune activation and metabolism with adverse events, haematology and biochemistry panels, genotype and physiological assessments

The investigators will biobank all samples for the duration of the BIOVACSAFE programme so that the investigators can selectively analyse different samples and different time points depending on the results generated, principally from the gene expression analysis of whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 18-45 years inclusive.
* Male: Female ratio - Screening will ensure that no more than 2/3 of the population should be of either male or female
* The subject is, in the opinion of the investigator: healthy based on medical history and clinical exam, with no active disease process that could interfere with the study endpoints.
* Has a body Mass Index ≥18 and ≤30
* Is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
* The subject has signed the ICF.
* The subject is available for follow-up for the duration of the study.
* The subject agrees to abstain from donating blood during their participation in the study, or longer if necessary.
* If the subject is a heterosexually active female, she is willing to use an effective method of contraception with partner (oral contraceptive pill; intrauterine device; injectable or implanted contraceptive; condoms incorporating spermicide if using these; physiological or anatomical sterility) from 30 days prior to, and 3 months after, vaccination. Willing to undergo urine pregnancy tests prior to vaccination at screening.
* The subject has venous access sufficient to allow blood sampling as per the protocol.

Exclusion Criteria:

* Pregnant or lactating at any point during the study from screening to final follow up.
* Hypersensitivity to the active components of FLUAD, any of the excipients, eggs, chicken proteins, kanamycin and neomycin sulphate, formaldehyde, and cetyltrimetholammonium bromide or those who have had a previous life-threatening reaction to previous influenza vaccinations.
* Presence of primary or acquired immunodeficiency states with a total lymphocyte count less than 1,200 per mm3 or presenting other evidence of lack of cellular immune competence e.g. leukaemias, lymphomas, blood dyscrasias, or patients receiving immunosuppressive therapy (including regular use of oral or parenteral corticosteroids).
* Use of any immune suppressing or immunomodulating drugs within 6 months of Visit 1.
* Regular use of non-steroidal anti-inflammatory drugs (oral or parenteral route) within 6 months of Visit 1 considered by the study physician as likely to interfere with immune responses.
* Current intake of excessive amounts of alcohol and/or caffeine (as evaluated by the investigator) and not willing to adapt this use during the study period.
* Currently performing extreme physical activities (as evaluated by the investigator) and not willing to adapt this use during the study period.
* Receipt of a vaccine within 30 days of visit 1, or requirement to receive another vaccine within the study period.
* Vaccination with the 2014/2015 seasonal influenza vaccine and/or any other seasonal influenza vaccine within the last 6 months before the first study visit.
* Presence of an acute severe febrile illness at time of immunisation.
* History of alcohol, narcotic, benzodiazepine, rilatine, or other substance abuse or dependence within the 12 months preceding Visit 1.
* Currently participating in another clinical study with an investigational or non-investigational drug or device, or has participated in a clinical trial within the 3 months preceding Visit 1.
* Any condition that, in the investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
* Receipt of blood products or immunoglobin, or blood donation, within 3 months of screening.
* Unable to read and speak Dutch or English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Frequency of local and systemic vaccine-related clinical events. | At all time points from vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in pulse. | At all time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in haematology (blood counts and ESR) parameters. | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in global gene expression measured on whole blood samples. | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in metabolic gene expression and pathway activation measured on whole blood samples. | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in serum HAI titre in serum samples. | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation values of adaptive cellular immune response via enumeration of HA-specific CD4+ T cells expressing activation markers and/or cytokines following in vitro stimulation and analysis by flow cytometry | At 7 days after vaccination
Change from pre-immunisation baseline values in concentration of selected cytokines and acute phase proteins in serum samples | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in PBMC cytokine secretion, proliferation or surface markers in response to in vitro antigen stimulation. | At selected time points from time of vaccination up to 28 days after vaccination
Genetic testing of subject (only when deemed necessary: may be SNIP analysis or full genome analysis) | Up to 2 years after vaccination
Change from pre-immunisation baseline values in body temperature. | At all time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in blood pressure. | At all time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in creatinin | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in CRP | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in AST/ALT | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in albumin | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in eGFR | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in GGT | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in total protein | At selected time points from time of vaccination up to 28 days after vaccination
Change from pre-immunisation baseline values in total prothrombin/fibrinogen | At selected time points from time of vaccination up to 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, Prof,MD, Principal Investigator — Center for Vaccinology
Locations (1):
- Center for Vaccinology, Ghent, East-Flanders, Belgium

REFERENCES:
- [Derived] Muturi-Kioi V, Lewis D, Launay O, Leroux-Roels G, Anemona A, Loulergue P, Bodinham CL, Aerssens A, Groth N, Saul A, Podda A. Neutropenia as an Adverse Event following Vaccination: Results from Randomized Clinical Trials in Healthy Adults and Systematic Review. PLoS One. 2016 Aug 4;11(8):e0157385. doi: 10.1371/journal.pone.0157385. eCollection 2016. PMID 27490698